CLINICAL TRIAL: NCT07325500
Title: Incretin Microdosing for Cardiometabolic Health in People With HIV: The REINFORCE Trial
Brief Title: Incretin Microdosing for Cardiometabolic Health in People With HIV
Acronym: REINFORCE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Colorado Denver - Anschutz Medical Campus (UCD-AMC) (Unknown); Massachusetts General Hospital (MGH) (Unknown)
Responsible Party: Principal Investigator, Jordan Elizabeth Lake, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-25-0376; 1R01DK142171-01A1 (NIH)
Record Dates: First submitted 2026-01-06; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Weight Gain
Keywords: semaglutide; HIV; obesity
MeSH Terms: conditions — Weight Gain; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose escalation to 2 mg semaglutide weekly then semaglutide microdosing at 0.5 mg weekly (Experimental): Participants will initiate semaglutide at 0.25 milligrams (mg) subcutaneously per week with dose titration up to 2.0 mg subcutaneously per week, over a total of 12 weeks. Dose titration will occur as follows: 0.25 mg weekly for 2 weeks, then 0.5 mg weekly for 2 weeks, then 1 mg weekly for 4 weeks, then 2.0 mg weekly for 4 weeks. Then, participants in this arm will receive microdosing with semaglutide at 0.5 mg subcutaneously every week during weeks 13-60.
  Interventions: Drug: Dose escalation to 2 mg semaglutide weekly then semaglutide microdosing at 0.5 mg weekly
- Dose escalation to 2 mg semaglutide weekly then no semaglutide (Experimental): Participants will initiate semaglutide at 0.25 milligrams (mg) subcutaneously per week with dose titration up to 2.0 mg subcutaneously per week, over a total of 12 weeks. Dose titration will occur as follows: 0.25 mg weekly for 2 weeks, then 0.5 mg weekly for 2 weeks, then 1 mg weekly for 4 weeks, then 2.0 mg weekly for 4 weeks. Then, participants in this arm will receive no semaglutide during weeks 13-60.
  Interventions: Drug: Dose escalation to 2 mg semaglutide weekly then no semaglutide

INTERVENTIONS:
Drug: Dose escalation to 2 mg semaglutide weekly then semaglutide microdosing at 0.5 mg weekly — Participants will initiate semaglutide at 0.25 milligrams (mg) subcutaneously per week with dose titration up to 2.0 mg subcutaneously per week, over a total of 12 weeks. Dose titration will occur as follows: 0.25 mg weekly for 2 weeks, then 0.5 mg weekly for 2 weeks, then 1 mg weekly for 4 weeks, then 2.0 mg weekly for 4 weeks. Then, participants in this arm will receive microdosing with semaglutide at 0.5 mg subcutaneously every week during weeks 13-60.
  Arms: Dose escalation to 2 mg semaglutide weekly then semaglutide microdosing at 0.5 mg weekly
Drug: Dose escalation to 2 mg semaglutide weekly then no semaglutide — Participants will initiate semaglutide at 0.25 milligrams (mg) subcutaneously per week with dose titration up to 2.0 mg subcutaneously per week, over a total of 12 weeks. Dose titration will occur as follows: 0.25 mg weekly for 2 weeks, then 0.5 mg weekly for 2 weeks, then 1 mg weekly for 4 weeks, then 2.0 mg weekly for 4 weeks. Then, participants in this arm will receive no semaglutide during weeks 13-60.
  Arms: Dose escalation to 2 mg semaglutide weekly then no semaglutide

SUMMARY:
The objectives of this study are as follows:

Primary Objective

* To determine the rate of weight regain in people living with human immunodeficiency virus (HIV) (PWH) receiving semaglutide microdosing vs. no additional drug following induction therapy.

Secondary Objectives

* To evaluate the tolerability of semaglutide microdosing in adults with HIV.
* To evaluate changes in weight, waist circumference (WC) and body mass index (BMI) over 12 weeks (W) of semaglutide weight loss induction and 48 W of semaglutide microdosing therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed human immunodeficiency virus type 1 (HIV-1)
* On antiretroviral therapy (ART) for greater than or equal to 24 weeks prior to entry and no change in regimen in the 12 weeks prior to entry or planned change for the study duration
* HIV-1 ribonucleic acid (RNA) <200 copies/mL at screening
* BMI greater than or equal to 30 kg/m2 or greater than or equal to 27 kg/m2 if also with greater than or equal to 1 weight-related comorbidity
* If taking anti-inflammatory or blood-pressure-/lipid-/glucose-lowering medications, no change in dose for greater than or equal to 12 weeks prior to entry and no plans to dose escalate for the study duration
* All participants must be willing and able to provide written informed consent and undergo all required study procedures

Exclusion Criteria:

* Weight greater than or equal to 400 pounds [due to dual X-ray absorptiometry (DXA) machine limitations] or unexplained weight change greater than or equal to 5% in the 12 weeks prior to entry
* Diagnosis of or on treatment for diabetes mellitus (stable metformin dosing for pre-diabetes not excluded)
* Current or planned use of medications for the treatment of obesity, or medications likely to cause significant changes in weight, during the study period
* Plans to newly engage in formal, intensive physical activity or diet (such as ketogenic or very low carbohydrate) programs during the study period
* Active eating disorder
* Use of human growth hormone, tesamorelin or anabolic steroids <12 weeks prior to entry, unless on a stable dose for >24 weeks prior to entry, or plans to start any of these medications while on study
* Active, severe delayed gastric emptying
* Prior bariatric surgery or major gastric surgery or plans for weight reduction surgery while on study
* Known retinopathy
* Personal or first-degree relative history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
* Untreated, poorly controlled or previously undiagnosed thyroid disease
* Chronic pancreatitis
* Known allergy/sensitivity to Glucagon-Like Peptide-1 Receptor Agonist (GLP-1RA)
* Poorly controlled or previously undiagnosed thyroid disease, defined as thyroid-stimulating hormone (TSH) <0.5 or >10 milli-international units per liter (mIU/L) at screening
* Active drug or alcohol use that, in the opinion of the investigator, would interfere with adherence to study requirements
* Pregnancy, nursing or plans for either during the study period
* Use of planned use of any immunomodulatory therapy HIV vaccine, investigational therapy or tumor necrosis factor (TNF-α) therapy during the study period
* Current serious illness requiring systemic treatment and/or hospitalization, in the opinion of site investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent weight regain from weeks 12-60 (microdosing period) | from week 12 to week 60
  The percent weight regain from weeks 12-60 (microdosing period), calculated as the median within-person: change in weight (kg) from weeks 60-12 (microdosing period) divided by the change in weight (kg) from weeks 12-0 (dose escalation period).

SECONDARY OUTCOMES:
Tolerability of semaglutide microdosing in participants as indicated by total number of serious adverse events (SAEs) and adverse events (AEs) | From baseline through week 60
  Total number of serious adverse events (SAEs) and adverse events (AEs) will be reported.
Absolute change in weight | Baseline, 12 weeks, 60 weeks
Percent change in weight | Baseline, 12 weeks, 60 weeks
Absolute change in body mass index (BMI) | Baseline, 12 weeks, 60 weeks
Percent change in body mass index (BMI) | Baseline, 12 weeks, 60 weeks
Absolute change in minimum waist circumference | Baseline, 12 weeks, 60 weeks
Percent change in minimum waist circumference | Baseline, 12 weeks, 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Lake, MD, MSc, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No